CLINICAL TRIAL: NCT00241644
Title: Multi-Center Study to Assess the Efficacy, Safety and Immunogenicity of 2 or 3 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine Given Concomitantly With Routine EPI Vaccinations in Healthy Infants
Brief Title: Vaccine Efficacy Against Rotavirus Diarrhea; Vaccine Given With Routine Childhood Vaccinations in Healthy African Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 102248; NCT00598468 (obsolete NCT alias)
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Rotavirus
Keywords: Rotavirus gastroenteritis; HRV vaccine
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Rotarix 3-Dose Group (Experimental): Subjects received 3 doses of Rotarix™ vaccine given concomitantly with routine EPI vaccines.
  Interventions: Biological: Rotarix™
- Rotarix 2-Dose Group (Experimental): Subjects received 1 dose of placebo followed by 2 doses of Rotarix™ vaccine given concomitantly with routine EPI vaccines.
  Interventions: Biological: Rotarix™; Biological: Placebo
- Placebo Group (Placebo Comparator): Subjects received 3 doses of placebo given concomitantly with routine EPI vaccines.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix™ — Two or Three doses, oral administration
  Other Names: GSK Biologicals' HRV vaccine
  Arms: Rotarix 2-Dose Group; Rotarix 3-Dose Group
Biological: Placebo — One or three doses, oral administration.
  Arms: Placebo Group; Rotarix 2-Dose Group

SUMMARY:
The primary objective of this study is to determine if the GSK Biologicals' human rotavirus (HRV) vaccine (pooled HRV groups) given concomitantly with routine expanded program on immunisation (EPI) vaccinations can prevent severe rotavirus gastroenteritis (≥11 on the 20-point Vesikari scoring system [Ruuska, 1990]) caused by the circulating wild-type RV strains during the period from 2 weeks after the last dose of HRV vaccine or placebo until Visit 5.

The primary objective will be reached if the lower limit of the 95% confidence interval (CI) on vaccine efficacy is >0%.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The study will have three groups: Rotarix 3-Dose Group, Rotarix 2-Dose Group and Placebo Group. Three-dose immunisation will be administered in healthy infants at approximately 6, 10, and 14 weeks of age. Routine EPI vaccinations will be administered concomitantly with the study vaccines. This study will also evaluate immunogenicity and safety relative to the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female child between, and including, 5 and 10 weeks of age at the time of the first study vaccination.
* Written informed consent obtained from the parent or guardian of the subject who is of legal age
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* In South Africa, birth weight > 2000 grams or if weight unknown, gestation period > 36 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Planned administration of a vaccine not foreseen by the study protocol within 14 days before each dose of study vaccine(s) and ending 14 days after.
* Chronic administration (defined as more than 14 days) of immunosuppressants since birth.
* History of use of experimental rotavirus vaccine.
* Previous routine vaccination except Bacille Calmette-Guérin (BCG), hepatitis B virus (HBV) and oral poliovirus (OPV) vaccination at birth
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract, intussusception or other medical condition determined to be serious by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Gastroenteritis within 7 days preceding the first study vaccine administration
* Previous confirmed occurrence of rotavirus gastroenteritis (RV GE).
* A family history of congenital or hereditary immunodeficiency.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* History of any neurologic disorders or seizures.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.

Ages: 5 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2089 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Malawi (4):
  - GSK Investigational Site, Bangwe, Blantyre
  - GSK Investigational Site, Limbe, Blantyre
  - GSK Investigational Site, Ndirande, Blantyre
  - GSK Investigational Site, Zingwanga, Blantyre
- South Africa (9):
  - GSK Investigational Site, Brits
  - GSK Investigational Site, Diepkloof, Soweto
  - GSK Investigational Site, Diepsloot
  - GSK Investigational Site, Eldorado Park Ext 9, Soweto
  - GSK Investigational Site, Karenpark
  - GSK Investigational Site, Mamelodi
  - GSK Investigational Site, Mamelodi East
  - GSK Investigational Site, Shoshanguve
  - GSK Investigational Site, Tembisa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cunliffe N et al. Efficacy of human rotavirus vaccine RIX4414 in Africa during the first year of life. Abstract presented at the 27th Annual Meeting of the European Society for Paediatric Infectious Disease (ESPID), Brussels, Belgium, 9-13 June 2009.
- [Background] Cunliffe NA, Witte D, Ngwira BM, Todd S, Bostock NJ, Turner AM, Chimpeni P, Victor JC, Steele AD, Bouckenooghe A, Neuzil KM. Efficacy of human rotavirus vaccine against severe gastroenteritis in Malawian children in the first two years of life: a randomized, double-blind, placebo controlled trial. Vaccine. 2012 Apr 27;30 Suppl 1(0 1):A36-43. doi: 10.1016/j.vaccine.2011.09.120. PMID 22520135
- [Background] Cunliffe NA et al. Efficacy of Human Rotavirus Vaccine RIX4414 in Malawian Infants in the first two years of life. Abstract presented at the 6th African Rotavirus Symposium, Johannesburg, South Africa, 2-3 August 2010.
- [Background] Madhi SA, Cunliffe NA, Steele D, Witte D, Kirsten M, Louw C, Ngwira B, Victor JC, Gillard PH, Cheuvart BB, Han HH, Neuzil KM. Effect of human rotavirus vaccine on severe diarrhea in African infants. N Engl J Med. 2010 Jan 28;362(4):289-98. doi: 10.1056/NEJMoa0904797. PMID 20107214
- [Background] Madhi S et al. Efficacy of the human rotavirus vaccine RIX4414 against rotavirus G2P[4]/g8p[4] strains in South African infants. Abstract presented at the 6th world congress of the World Society for Pediatric Infectious Diseases (WSPID), Buenos Aires, Argentina, 18-22 November 2009.
- [Background] Madhi SA, Kirsten M, Louw C, Bos P, Aspinall S, Bouckenooghe A, Neuzil KM, Steele AD. Efficacy and immunogenicity of two or three dose rotavirus-vaccine regimen in South African children over two consecutive rotavirus-seasons: a randomized, double-blind, placebo-controlled trial. Vaccine. 2012 Apr 27;30 Suppl 1:A44-51. doi: 10.1016/j.vaccine.2011.08.080. PMID 22520136
- [Background] Nakagomi T, Nakagomi O, Dove W, Doan YH, Witte D, Ngwira B, Todd S, Duncan Steele A, Neuzil KM, Cunliffe NA. Molecular characterization of rotavirus strains detected during a clinical trial of a human rotavirus vaccine in Blantyre, Malawi. Vaccine. 2012 Apr 27;30 Suppl 1(0 1):A140-51. doi: 10.1016/j.vaccine.2011.09.119. PMID 22520123
- [Background] Neuzil K et al. Immunogenicity of human rotavirus vaccine RIX4414 in South African and Malawian infants. Abstract presented at the 6th world congress of the World Society for Pediatric Infectious Diseases (WSPID), Buenos Aires, Argentina, 18-22 November 2009.
- [Background] Neuzil K et al. RIX4414 is protective against severe RVGE caused by diverse rotavirus serotypes during the first year of life in African infants. Abstract presented at the 27th Annual Meeting of the European Society for Paediatric Infectious Disease (ESPID), Brussels, Belgium, 9-13 June 2009.
- [Background] Steele AD et al. Efficacy of human rotavirus vaccine, Rotarix™ against severe gastroenteritis caused by diverse circulating rotavirus strains in African infants. Abstract presented at the 7th World Congress for World Society for Pediatric Infectious Diseases (WSPID). Melbourne, Australia, 16-19 November 2011.
- [Background] Steele D et al. Diverse circulating rotavirus strains during the first year of life in African infants. Abstract presented at 10th International symposium on dsRNA Viruses, Hamilton Island, QLD, Australia, 21-25 June 2009.
- [Derived] Gruber JF, Becker-Dreps S, Hudgens MG, Brookhart MA, Thomas JC, Jonsson Funk M. Timing and predictors of severe rotavirus gastroenteritis among unvaccinated infants in low- and middle-income countries. Epidemiol Infect. 2018 Apr;146(6):698-704. doi: 10.1017/S0950268818000626. Epub 2018 Mar 22. PMID 29564996
- [Derived] Madhi SA, Cunliffe NA, Steele D, Witte D, Kirsten M, Louw C, Ngwira B, Victor JC, Gillard PH, Cheuvart BB, Han HH, Neuzil KM. Effect of human rotavirus vaccine on severe diarrhea in African infants. Malawi Med J. 2016 Sep;28(3):108-114. PMID 27895844
- [Derived] Steele AD, Neuzil KM, Cunliffe NA, Madhi SA, Bos P, Ngwira B, Witte D, Todd S, Louw C, Kirsten M, Aspinall S, Van Doorn LJ, Bouckenooghe A, Suryakiran PV, Han HH. Human rotavirus vaccine Rotarix provides protection against diverse circulating rotavirus strains in African infants: a randomized controlled trial. BMC Infect Dis. 2012 Sep 13;12:213. doi: 10.1186/1471-2334-12-213. PMID 22974466
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 102248 are summarised with study 111274 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only subjects from Malawi and from Cohort 2 South Africa were asked to continue the study for a second follow-up period (Year 2).
Pre-assignment Details: Of the total of 4941 subjects enrolled in this study, 2 subjects were allocated a subject number but did not get any study vaccine administered. Hence, only 4939 subjects were considered as 'started'.
  For the second follow-up period, as mentioned in the protocol the results are presented for Rotarix Pooled and Placebo Groups only.
Groups:
- Rotarix 2-dose Group: Subjects received 1 dose of placebo followed by 2 doses of Rotarix™ (rotavirus vaccine).
- Rotarix 3-dose Group: Subjects received 3 doses of Rotarix™ (rotavirus vaccine).
- Placebo Group: Subjects received 3 doses of placebo.
- Rotarix Pooled Group: Subjects received 2 or 3 doses of Rotarix™ (rotavirus vaccine).
Period: First Efficacy Period (Year 1)
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Placebo Group | Rotarix Pooled Group
Started | 1647 | 1651 | 1641 | 3298
Completed | 1420 | 1383 | 1392 | 2803
Not Completed | 227 | 268 | 249 | 495
Not completed — Adverse Event | 46 | 45 | 45 | 91
Not completed — Protocol Violation | 3 | 5 | 4 | 8
Not completed — Withdrawal by Subject | 59 | 74 | 81 | 133
Not completed — Lost to Follow-up | 116 | 142 | 116 | 258
Not completed — Non-compliance | 2 | 1 | 2 | 3
Not completed — Return dates not reliable | 1 | 0 | 0 | 1
Not completed — Vaccinated at regular clinic | 0 | 0 | 1 | 0
Not completed — Subject's parent passed away | 0 | 1 | 0 | 1
Period: Second Efficacy Period (Year 2)
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Placebo Group | Rotarix Pooled Group
Started | 771 | 754 | 746 | 1525
Completed | 710 | 697 | 682 | 1407
Not Completed | 61 | 57 | 64 | 118
Not completed — Adverse Event | 11 | 9 | 12 | 20
Not completed — Protocol Violation | 2 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 4 | 3 | 2 | 7
Not completed — Lost to Follow-up | 43 | 43 | 46 | 86
Not completed — Consenting parent passed away | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Placebo Group | Rotarix Pooled Group | Total
Number analyzed (Participants) | 1647 | 1651 | 1641 | 3298 | 8237
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 6.3 (0.92) | 6.4 (0.98) | 6.4 (0.97) | 6.4 (0.95) | 6.4 (0.95)
Gender [Count of Participants; unit: Participants]
  Female | 811 | 839 | 800 | 1650 | 4100
  Male | 836 | 812 | 841 | 1648 | 4137

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis (RV GE) Caused by the Circulating Wild-type Rotavirus Strain
Description: Number of subjects presenting with three or more looser than normal stools or watery stools within a day, occurring after administration of dose 1 of study vaccine in which rotavirus other than vaccine strain was identified in a stool sample with a score ≥ 11 on the 20-point Vesikari scoring system.
Time Frame: From 2 weeks after the last vaccine or placebo dose up to 1 year of age
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy
Measure: Number; unit: subjects
Groups:
- Rotarix Pooled Group: For some data analyses, the 2 Groups receiving Rotarix (Rotarix 2-dose Group & Rotarix 3-dose Group) were pooled into Rotarix pooled Group.
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1496 | 1478 | 2974 | 1443
subjects | 30 | 26 | 56 | 70

2. Secondary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis Caused by the Circulating Wild-type Rotavirus Strain, Classified by Rotavirus Type
Description: Number of subjects presenting with three or more looser than normal stools within a day, occurring after administration of dose 1 of study vaccine in which rotavirus other than vaccine strain was identified in a stool sample with a score ≥ 11 on the 20-point Vesikari scoring system.
  Rotavirus types were G1 wild type (WT) and non-G1.
Time Frame: From 2 weeks after the last vaccine or placebo dose up to 1 year of age
Population: Analysis was performed on the ATP cohort for efficacy
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1496 | 1478 | 2974 | 1443
subjects
  G1 WT | 8 | 9 | 17 | 23
  Non-G1 | 22 | 17 | 39 | 47

3. Secondary Outcome: Number of Subjects Reporting Any Rotavirus Gastroenteritis Caused by the Circulating Wild-type Rotavirus Strain
Description: Number of subjects presenting with three or more looser than normal stools or watery stools within a day, occurring after administration of dose 1 of study vaccine in which rotavirus other than vaccine strain was identified in a stool sample.
Time Frame: From 2 weeks after the last vaccine or placebo dose up to 1 year of age
Population: Analysis was performed on the ATP cohort for efficacy
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1496 | 1478 | 2974 | 1443
subjects | 93 | 74 | 167 | 174

4. Secondary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis Caused by the Circulating Wild-type Rotavirus Strain
Description: as for outcome 1
Time Frame: From the first vaccine or placebo dose up to 1 year of age
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1647 | 1651 | 3298 | 1641
subjects | 37 | 31 | 68 | 83

5. Secondary Outcome: In South Africa, Number of Subjects With Severe Rotavirus Gastroenteritis Caused by the Circulating Wild-type Rotavirus Strain
Description: as for outcome 1
Time Frame: From 2 weeks after the third dose of vaccine or placebo up to 1 year of age
Population: Analysis was performed on the ATP cohort for efficacy, only for the subset of subjects in South Africa who were fully vaccinated before the beginning of the rotavirus season.
  For this analysis, data from Rotarix 2-dose Group and Rotarix 3-dose Group were pooled into one group (Rotarix pooled Group).
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 478 | 468 | 946 | 468
subjects | 5 | 3 | 8 | 20

6. Secondary Outcome: Number of Subjects Reporting Severe Gastroenteritis of Any Cause
Description: Number of subjects with gastroenteritis (three or more looser than normal stools or watery stools within a day) that scored ≥ 11 on the 20-point Vesikari scoring system.
Time Frame: From 2 weeks after the last vaccine or placebo dose up to 1 year of age
Population: Analysis was performed on the ATP cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1496 | 1478 | 2974 | 1443
subjects | 134 | 122 | 256 | 178

7. Secondary Outcome: Number of Subjects Hospitalized and/or With Supervised Re-hydration Therapy Due to Rotavirus Gastroenteritis (RV GE) Caused by the Circulating Wild-type Rotavirus Strain
Description: RV GE caused by the circulating wild-type rotavirus strain: three or more looser than normal stools or watery stools within a day, occurring after administration of dose 1 of study vaccine in which rotavirus other than vaccine strain was identified in a stool sample collected as soon as possible after the symptoms begin.
Time Frame: From 2 weeks after the last vaccine or placebo dose up to 1 year of age
Population: Analysis was performed on the ATP cohort for efficacy
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1496 | 1478 | 2974 | 1443
subjects | 78 | 64 | 142 | 156

8. Secondary Outcome: For Subjects in Cohort 2 South Africa and the Cohort in Malawi: Number of Subjects With Severe Rotavirus Gastroenteritis (RV GE) Caused by the Circulating Wild-type Rotavirus Strains
Description: as for outcome 1
Time Frame: During the period from 2 weeks after the last dose of vaccine or placebo until study end
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for efficacy of the combined efficacy follow-up periods.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 1873 | 891
subjects |  |  | 81 | 66

9. Secondary Outcome: For Subjects in Cohort 2 South Africa and the Cohort in Malawi: Number of Subjects With Severe Rotavirus Gastroenteritis (RV GE) Caused by the Circulating Wild-type Rotavirus Strains
Description: as for outcome 1
Time Frame: During the period from 1 year of age to study end
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for efficacy of the second efficacy period.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 1500 | 712
subjects |  |  | 35 | 21

10. Secondary Outcome: For Subjects in Cohort 2 South Africa and the Cohort in Malawi: Number of Subjects Hospitalized and/or With Supervised Re-hydration Therapy Due to Rotavirus Gastroenteritis (RV GE) Episode Caused by the Circulating Wild-type RV Strains
Description: as for outcome 7
Time Frame: During the period from 2 weeks after the last dose of vaccine or placebo until study end
Population: The analysis was performed on the ATP cohort for efficacy of the combined efficacy follow-up periods.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 1873 | 891
subjects |  |  | 159 | 118

11. Secondary Outcome: For Subjects in Cohort 2 South Africa and the Cohort in Malawi: Number of Subjects Hospitalized and/or With Supervised Re-hydration Therapy Due to Rotavirus Gastroenteritis (RV GE) Episode Caused by the Circulating Wild-type RV Strains
Description: as for outcome 7
Time Frame: During the period from 1 year of age to study end
Population: The analysis was performed on the ATP cohort for efficacy of the second efficacy period.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 1500 | 712
subjects |  |  | 58 | 26

12. Secondary Outcome: For Subjects in Cohort 2 South Africa and the Cohort in Malawi: Number of Subjects With Severe Rotavirus Gastroenteritis Caused by the Circulating Wild-type Rotavirus Strains, Classified by Rotavirus Type
Description: Number of subjects presenting with three or more looser than normal stools or watery stools within a day, occurring after administration of dose 1 of study vaccine in which rotavirus other than vaccine strain was identified in a stool sample with a score ≥ 11 on the 20-point Vesikari scoring system.
  Rotavirus types were G1 wild type (WT) and non-G1.
Time Frame: During the period from 2 weeks after the last dose of vaccine or placebo until study end
Population: The analysis was performed on the ATP cohort for efficacy of the combined efficacy follow-up periods.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 1873 | 891
subjects
  G1 WT |  |  | 21 | 20
  Non-G1 |  |  | 60 | 48

13. Secondary Outcome: For Subjects in Cohort 2 South Africa and the Cohort in Malawi: Number of Subjects With Severe Rotavirus Gastroenteritis Caused by the Circulating Wild-type Rotavirus Strains, Classified by Rotavirus Type
Description: as for outcome 12
Time Frame: During the period from 1 year of age to study end
Population: The analysis was performed on the ATP cohort for efficacy of the second efficacy period.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 1500 | 712
subjects
  G1 WT |  |  | 10 | 11
  Non-G1 |  |  | 25 | 10

14. Secondary Outcome: Number of Subjects With Adverse Events (AEs) or Serious Adverse Events (SAEs) Leading to Drop Out
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From the first dose of vaccine or placebo up to end of the study
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1647 | 1651 | 3298 | 1641
subjects | 57 | 54 | 111 | 56

15. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From the first dose of vaccine or placebo up to end of the study
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1647 | 1651 | 3298 | 1641
subjects | 222 | 199 | 421 | 246

16. Secondary Outcome: Geometric Mean Concentration of Anti-rotavirus Immunoglobulin A (IgA) Antibodies in Initially Seronegative Subjects
Description: An initially seronegative subject is a subject whose IgA antibody concentration was below the assay cut-off value of 20 Units per milliliter (U/mL) before administration of the first vaccine dose.
Time Frame: One month after the last vaccine dose
Population: Analysis was performed on the ATP cohort for immunogenicity, only for initially seronegative subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter (U/mL)
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 106 | 115 | 221 | 111
Units per milliliter (U/mL) | 56.6 [38.9 to 82.3] | 79.4 [54.7 to 115.2] | 67.5 [51.9 to 87.8] | 23.4 [16.8 to 32.5]

17. Secondary Outcome: Number of Seroconverted Subjects
Description: Seroconverted subjects are defined as subjects with appearance of anti-rotavirus IgA antibody concentration ≥ 20 U/mL in subjects initially (i.e. prior to the first dose of vaccine or placebo) seronegative for rotavirus.
Time Frame: One month after the last vaccine or placebo dose
Population: Analysis was performed on the ATP cohort for immunogenicity, only for inititally seronegative subjects.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 106 | 115 | 221 | 111
subjects | 57 | 72 | 129 | 25

18. Secondary Outcome: Geometric Mean Concentration of Anti-rotavirus Immunoglobulin A (IgA) Antibodies
Description: Geometric mean concentrations are given as Units per milliliter (U/mL).
Time Frame: One month after the last vaccine or placebo dose
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1160 | 1138 | 2298 | 1125
U/mL | 72.5 [65.2 to 80.6] | 67.9 [60.8 to 75.9] | 70.2 [65.0 to 75.8] | 21.8 [19.8 to 24.0]

19. Secondary Outcome: Number of Seropositive Subjects
Description: Seropositive subjects are defined as subjects with anti-rotavirus IgA antibody concentration ≥ 20 U/mL.
Time Frame: One month after the last vaccine or placebo dose
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Number analyzed (Participants) | 1160 | 1138 | 2298 | 1125
subjects | 756 | 706 | 1462 | 262

ADVERSE EVENTS:
Arm/Group | Rotarix 2-dose Group | Rotarix 3-dose Group | Rotarix Pooled Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 222/1647 | 199/1651 | 421/3298 | 246/1641
Other Adverse Events (participants affected / at risk) | 0/1647 | 0/1651 | 0/3298 | 0/1641
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix 2-dose Group (N=1647) | Rotarix 3-dose Group (N=1651) | Rotarix Pooled Group (N=3298) | Placebo Group (N=1641)
Gastroenteritis (Infections and infestations) | 94 | 67 | 161 | 104
Pneumonia (Infections and infestations) | 55 | 54 | 109 | 64
Bronchopneumonia (Infections and infestations) | 29 | 25 | 54 | 25
Sepsis (Infections and infestations) | 33 | 28 | 61 | 29
Bronchiolitis (Infections and infestations) | 21 | 17 | 38 | 17
Malaria (Infections and infestations) | 19 | 25 | 44 | 33
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 14 | 1
Meningitis (Infections and infestations) | 7 | 4 | 11 | 2
Pneumocystis jiroveci pneumonia (Infections and infestations) | 4 | 4 | 8 | 5
Febrile convulsion (Nervous system disorders) | 4 | 7 | 11 | 6
Anemia (Blood and lymphatic system disorders) | 2 | 6 | 8 | 2
Pulmonary tuberculosis (Infections and infestations) | 3 | 3 | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 6 | 2
Kwashiorkor (Metabolism and nutrition disorders) | 3 | 4 | 7 | 8
Gastrointestinal disorder (Gastrointestinal disorders) | 4 | 2 | 6 | 3
Malnutrition (Metabolism and nutrition disorders) | 5 | 0 | 5 | 1
Death (General disorders) | 2 | 2 | 4 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 3
Oral candidiasis (Infections and infestations) | 2 | 1 | 3 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 2 | 2
Pneumonia viral (Infections and infestations) | 3 | 0 | 3 | 2
Pyrexia (General disorders) | 1 | 3 | 4 | 4
Sudden infant death syndrome (General disorders) | 0 | 2 | 2 | 2
Croup infectious (Infections and infestations) | 1 | 1 | 2 | 1
Marasmus (Metabolism and nutrition disorders) | 3 | 5 | 8 | 4
Otitis media (Infections and infestations) | 2 | 1 | 3 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1 | 2 | 0
Encephalitis (Nervous system disorders) | 1 | 0 | 1 | 2
Heart disease congenital (Congenital, familial and genetic disorders) | 1 | 1 | 2 | 0
Ileus paralytic (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 2 | 2 | 2
Otitis media acute (Infections and infestations) | 1 | 1 | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0
Status epilepticus (Nervous system disorders) | 1 | 1 | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 2
Tonsillitis (Infections and infestations) | 2 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 2
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 1 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 2 | 3 | 3
Fontanelle bulging (Nervous system disorders) | 0 | 1 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 3
Staphylococcal skin infection (Infections and infestations) | 1 | 1 | 2 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 4 | 6 | 4
Abscess (Infections and infestations) | 0 | 1 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 1 | 0
Adenoidectomy (Surgical and medical procedures) | 1 | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Blindness (Eye disorders) | 1 | 0 | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0
Cerebral malaria (Infections and infestations) | 1 | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 1 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 1 | 0
Fractured skull depressed (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypovolaemic shock (Cardiac disorders) | 0 | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Klebsiella bacteremia (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Parotid abscess (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 2 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis neonatal (Infections and infestations) | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 1 | 2 | 0
Varicella (Infections and infestations) | 1 | 0 | 1 | 0
Viral tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 2
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Immunosuppression (Immune system disorders) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Perianal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Keratitis herpetic (Infections and infestations) | 1 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 1 | 0
Salmonella sepsis (Infections and infestations) | 0 | 1 | 1 | 0
skin infection (Infections and infestations) | 0 | 1 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.